CLINICAL TRIAL: NCT05854225
Title: Thiotepa Incorporating TBI/Cy Conditioning Regimen Followed by HSCT for EBV-HLH With Central Nervous System Involvement: a Prospective Single-arm Clinical Study
Brief Title: Thiotepa Incorporating TBI/Cy Conditioning Regimen for EBV-HLH With Central Nervous System Involvement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhao Wang, Professor and Head of hematology, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-P2-250-01
Record Dates: First submitted 2023-04-20; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: HLH
MeSH Terms: interventions — Thiotepa

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single-arm (Other): a prospective single-arm clinical study
  Interventions: Drug: Thiotepa

INTERVENTIONS:
Drug: Thiotepa — Thiotepa is an alkylating agent that is routinely used in solid tumors, but it is able to cross the blood-brain barrier into the center.
  Other Names: TT

SUMMARY:
EBV-HLH is the most common in virus-associated hemophagocytic syndrome (VAHS). There are no uniform clinical criteria for the diagnosis of CNS-HLH. And there is still a lack of international consensus on the treatment for CNS-HLH. Following allogeneic HSCT after HLH induction therapy is recommended for CNS-HLH. One of the major factors influencing the transplantation effect is conditioning. Therefore, we conduct a prospective clinical study to explore the efficacy and safety of thiotepa incorporating TBI/Cy conditioning regimen followed by allogeneic hematopoietic stem cell transplantation for EBV-HLH with central nervous system involvement.

DETAILED DESCRIPTION:
HLH is an immune disorder characterized by a potentially fatal cytokine storm induced by uncontrolled T lymphocyte and macrophage activation. EBV-HLH is the most common in virus-associated hemophagocytic syndrome (VAHS). There are no uniform clinical criteria for the diagnosis of CNS-HLH. And there is still a lack of international consensus on the treatment for CNS-HLH. CNS involvement is one of the factors in the poor prognosis for HLH. Following allogeneic HSCT after HLH induction therapy is recommended for CNS-HLH. One of the major factors influencing the transplantation effect is conditioning. Therefore, we conduct a prospective clinical study to explore the efficacy and safety of thiotepa incorporating TBI/Cy conditioning regimen followed by allogeneic hematopoietic stem cell transplantation for EBV-HLH with central nervous system involvement.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as HLH according to HLH-04 diagnostic criteria.
2. a significant increase of EBV-DNA copies/ml in peripheral blood or tissue or EBER(+) in tissue specimens or peripheral blood.
3. Cerebrospinal fluid EBV-DNA ≥5×10^2 copies/ml.
4. Estimated survival time ≥ 1 month.
5. Age 18~60， gender is not limited.
6. Total bilirubin ≤ 2 times the upper limit of normal; serum creatinine ≤ normal value before study entry.
7. Serum HIV antigen or antibody negative.
8. HCV antibody negative.
9. HBsAg negative, HBcAb negative. If any of the above is positive, then HBV-DNA titer in peripheral blood is required less than 1×102 copies/ml before enrollment.
10. Cardiac ultrasound LVEF≥50%.
11. Women in the child-bearing period must not be pregnant as determined by a pregnancy test and must be willing to use effective contraception during the trial and for ≥ 12 months after the last dose. Pregnant and lactating women cannot participate. All male subjects accept contraception during the trial and for ≥6 months after the last dose.
12. Signed informed consent.

Exclusion Criteria:

1. Heart function above grade II (NYHA).
2. Active bleeding of the internal organs(digestive tract, lung, brain, etc.).
3. Uncontrolled infection (pulmonary infection, intestinal infection, etc.).
4. Severe mental illness.
5. Patients are unable to comply during the trial and/or follow-up phase.
6. Participate in other clinical research at the same time.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
The clinical remission rate | 24 weeks
  The number of cases with complete response (CR) and partial response (PR) after transplantation as a percentage of the total cases.

CONTACTS AND LOCATIONS:
Overall Officials: wang zhao, MD, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China